CLINICAL TRIAL: NCT06749132
Title: Deep Learning-enhanced Personalized Monitoring of Aortic Stenosis - The DETECT-AS Prognostic Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Icahn School of Medicine at Mount Sinai (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2000038730; R01AG089981 (NIH)
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; artificial intelligence
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiogram — All study participants will undergo a clinical transthoracic echocardiogram (TTE) performed by certified echocardiography technicians. The TTE includes standard transthoracic examination with acquisition of B-mode, color and spectral Doppler images and videos in line with standard echocardiographic guidelines.

SUMMARY:
This study will evaluate the validity of a digital biomarker score for precision risk stratification among older adults with aortic sclerosis or mild aortic stenosis (AS) at three US health systems.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or older
2. Prior transthoracic echocardiogram within the past 2-3 years showing aortic sclerosis without stenosis or mild AS

Exclusion Criteria:

1. Opted out of research studies
2. Non-English speaking
3. Any echocardiogram within 24 months of medical record review.
4. Prior history of aortic valve replacement or repair, including transcatheter and surgical AVR with either a bioprosthetic or mechanical valve
5. Presence of implantable cardiac devices, including permanent cardiac pacer, implantable cardioverter-defibrillator, or left ventricular assist device
6. Prior heart transplant
7. History of dementia
8. Unable to attend study visit at echocardiogram lab within four years of most recent echocardiogram.
9. Documented life expectancy of <1 year or current participation in hospice services

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: US adults aged 65 and older with an echocardiogram within the prior 2-3 years that showed aortic sclerosis without stenosis or mild aortic stenosis (AS).
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Annualized change in AV Vmax in m/sec/years | From baseline TTE to TTE performed at enrollment
  The primary outcome measure is the annualized change in AV Vmax in m/sec/years, defined as the absolute difference between the value on the enrollment and baseline echocardiogram measurement, divided by the time difference between the studies.

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Khera, MD, MS, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale New Haven Health System, New Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Methodist Hospital Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available following publication of primary results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code